CLINICAL TRIAL: NCT00312078
Title: Effect of Yogurt Supplementation on Psychometric Test Performance in Cirrhotic Patients With Minimal Hepatic Encephalopathy. A Prospective Pilot Trial.
Brief Title: Effect of Yogurt on Minimal Hepatic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCRC protocol 810; HRRC 360-05
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Cirrhosis; Minimal Hepatic Encephalopathy
Keywords: Minimal Hepatic Encephalopathy; Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Yogurt Supplementation

SUMMARY:
The purpose of this study is to determine whether a special yogurt can improve performance on certain tests of intelligence and decrease liver inflammation in patients with cirrhosis.

DETAILED DESCRIPTION:
Introduction: Cirrhosis is one of the leading causes of death in the United States. Minimal hepatic encephalopathy (MHE) is a significant complication of cirrhosis, which is often not treated because of perceived subclinical nature of this condition and the adverse effects and expense of available medications such as lactulose or rifaximin. There is evidence that small intestinal bacterial overgrowth can contribute to the development of MHE and cirrhosis in murine and human studies. Probiotics are live bacteria that can modify the indigenous intestinal bacterial flora and have been recently used in the treatment of hepatic encephalopathy in patients with cirrhosis.

Our aim is to evaluate the effect of probiotic supplementation via yogurt on liver function and inflammatory markers of bacterial translocation and psychometric test performance in cirrhotic patients with MHE in a prospective pilot trial.

Methods: 30 patients with MHE 2:1 i.e. 20 will be randomized into supplementation with yogurt to be taken 6 ounces twice a day for 60 days and 10 patients will be followed up without yogurt supplementation. All patients will undergo liver function tests, basic metabolic panel, INR, venous ammonia, IL-6 and TNF-alpha at baseline, 30 days and at 60 days. All patients will also undergo psychometric testing with number connection test A, digit symbol test, block design and inhibitory control test at baseline and 60 days. Regular questioning about adherence to yogurt. Collection of yogurt tops as proof of yogurt consumption and review of intake diary will be done at 30 and 60 days from patients randomized to yogurt supplementation.

Importance: There has been only one human study on the modification of gut flora as a therapeutic tool for improvement of MHE in cirrhosis, however that study included alcoholic liver disease and comprised of Chinese patients, therefore etiologies of liver diseases studied were different from those predominant in the United States. Since MHE can adversely affect quality of life and overall prognosis, simple, targeted therapies are needed to treat it. We believe that our pilot study will help delineate human gut flora as a definite target for therapy of cirrhosis and MHE and pave the way for future large-scale studies on this subject.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis diagnosed on clinical grounds (within 3 months of enrollment)
* MHE diagnosed by abnormalities in a psychometric battery (NCT-A,BDT,DST and ICT)

Exclusion criteria:

* Current or recent (< 6 month) use of alcohol
* Co-existing cause of liver dysfunction
* Use of antibiotics within last 6 weeks
* Infection or gastrointestinal hemorrhage within the last 6 weeks
* Hepatocellular carcinoma
* Psychoactive drug use, including interferon concurrently

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Reversal of minimal hepatic encephalopathy

SECONDARY OUTCOMES:
Decrease in AST/ALT

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan S Bajaj, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- GCRC Medical College of Wisconsin, Milwaukee, Wisconsin, United States